CLINICAL TRIAL: NCT06351007
Title: Effect of an Educational Program on Dietary Adherence, Nutritional Knowledge, Nutritional Status, Metabolic Control and Quality of Life in Predialysis, Peritoneal Dialysis and Hemodialysis Patients With Chronic Kidney Disease
Brief Title: Educational Program on Dietary Adherence and Nutritional Knowledge in Chronic Kidney Disease Patients (EPAK)
Acronym: EPAK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMM-4650-23-24-1
Record Dates: First submitted 2024-03-07; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-01

CONDITIONS: Chronic Kidney Disease; Predialysis; Peritoneal Dialysis; Hemodialysis; Educational Activities; Adherence; Nutritional Status
Keywords: Education program; Adherence; Nutritional knowledge; Nutritional status; Quality of Life; Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Psychosocial Intervention; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): The control group will consist of both pre-dialysis and dialysis patients.They will receive standard nutritional care consisting of dietary prescription with follow-up for questions and adjustment of the meal plan every 2 months.
  Interventions: Other: Standard care
- Intervention predialysis (Experimental): This group will consist of pre-dialysis patients in Kidney Disease Improving Global Outcomes (KDIGO) stages 3 to 5 who will receive, in addition to the meal plan, a nutritional education program with psychological support.The meal plan will have the same characteristics as in the control group.
  The educational program will have a duration of 5 monthly sessions . Simultaneously, monthly sessions will be held in groups of 5 patients, with a group of clinical psychologists.
  Interventions: Other: Nutritional education and psychological intervention
- Intervention dialysis (Experimental): This group will consist of peritoneal dialysis and hemodialysis patients who will receive, in addition to the meal plan, a nutritional education program with psychological support.The meal plan will have the same characteristics as in the control group.
  The educational program will have a duration of 5 monthly sessions . Simultaneously, monthly sessions will be held in groups of 5 patients, with a group of clinical psychologists.
  Interventions: Other: Nutritional education and psychological intervention

INTERVENTIONS:
Other: Nutritional education and psychological intervention — In the two intervention groups, after the delivery of the meal plan, the educational and psychological intervention will begin, with a duration of 5 months. The main objective of the educational program in pre-dialysis patients is to delay the progression of renal damage and in dialysis patients is control of complications. The content of monthly educational sessions will be:
  Month 1: proteins (predialysis group), potassium (dialysis group) Month 2: Sodium and fluids (predialysis group), phosphorus (dialysis group) Month 3: Phosphorus (predialysis group), sodium and fluids (dialysis group) Month 4: Potassium (predialysis group), proteins (dialysis group) Month 5: Myths and facts about food (both groups) Simultaneously, group psychological sessions will be carried out, aimed at modifying patient behaviors to increase adherence to diet plan through understanding the patient´s situation, promoting the development of healthy behaviors, barrier identification and goal setting
  Arms: Intervention dialysis; Intervention predialysis
Other: Standard care — The control group (predialysis and dialysis patients) will receive standard nutritional care consisting of dietary prescription with follow-up for questions and adjustment of the meal plan every 2 months.
  Based on the nutritional status, biochemical parameters and stage of renal disease, the meal plan will be calculated.
  The characteristics of the diet will be as follows:
  Calories - 30 kcal/Kg ideal body weight/day Protein - 0.8 g/kg ideal body weight/day (predialysis group) 1.2 kg ideal body weight/day (dialysis group) Carbohydrates - 50-60% of total calorie content Lipids - 30% of total calorie content Sodium < 2300 mg/day Potassium < 2000 mg/day Phosphorus < 1000 mg/day Fluids - Urine output + 500 ml
  Arms: Control

SUMMARY:
A fundamental strategy to improve adherence to nutritional treatment in patients with chronic kidney disease is the implementation of educational programs. The aim of this study is to evaluate the effect of a multidisciplinary educational program on dietary adherence, nutritional knowledge, nutritional status, metabolic control and quality of life in patients with chronic kidney disease, predialysis, peritoneal dialysis and hemodialysis.

A randomized clinical trial will be carried out, in which patients who meet the inclusion criteria will be randomly assigned to three possible groups: predialysis educational intervention, dialysis educational intervention and control group. At the initial visit, the nutritional status will be evaluated by means of anthropometric parameters, screening and dynamometry, the biochemical parameters of interest will be extracted from the clinical record, nutritional knowledge and quality of life will be evaluated, and the diet will be explained. In the second visit, adherence to the diet will be evaluated and the food registry will be carried out. In the intervention groups, the educational program will begin with a duration of five months. Patients will come twice a month to the hospital to participate in the educational sessions and attend group psychology sessions. After completion of the educational program, the same measurements as at the beginning of the study will be carried out in the three groups.

DETAILED DESCRIPTION:
Nutritional treatment is of great importance for an adequate control of chronic kidney disease. An adequate and personalized design of the nutritional plan, as well as permanent follow-up and support, allow slowing down the evolution of the disease, preserving the nutritional status, improving survival expectations, as well as the patient's quality of life. A difficulty faced by the health team dedicated to the management of chronic kidney disease (CKD) is the poor adherence of patients to treatment, specifically to nutritional therapy. Many patients with CKD express that adherence to dietary restrictions is the most difficult part of the treatment regimen because it affects food preferences and alters lifestyle. Approximately, only 31.5% of patients have adequate dietary adherence.

Educational programs increase knowledge about CKD and renal nutrition, improve concentrations of biochemical parameters, and improve quality of life; however, it is not clear that they improve adherence to the dietary plan. Although knowledge is a necessary precondition for behavioral change, it is not sufficient to improve adherence to treatment. In this regard, psychological interventions, designed to increase patients' confidence and self-management by increasing skills and strategies for behavioral change, can be useful to improve metabolic control and adherence. Given the above, it is essential to design and implement multidisciplinary educational interventions to improve patients' adherence to treatment.

The aim of the study is to evaluate the effect of a multidisciplinary educational program on dietary adherence, nutritional knowledge, nutritional status, metabolic control and quality of life in patients with chronic kidney disease, predialysis, peritoneal dialysis and hemodialysis.

The study subjects will be active patients of the nephrology clinic of the National Institute of Medical Science and Nutrition, who meet the inclusion criteria. They will be invited to participate in the protocol and those who accept will sign the informed consent form. Thirty-two pre-dialysis patients will be recruited, of whom 21 will receive the educational intervention and 11 will be part of the control group. Similarly, 32 dialysis patients (peritoneal or hemodialysis) will be recruited, 21 of whom will receive the educational intervention and 11 will be part of the control group.The sample size was estimated through the comparison of means with the analysis of variance formula for three groups, based on the main variable of the study, which is dietary adherence. A confidence level of 95%, statistical power of 80% and losses of 30% were taken into account.

After recruitment and signature of the consent form, the three study groups were formed by block randomization: control group, group of pre-dialysis patients and group of dialysis patients.

The following variables will be extracted from the clinical record: age, sex, educational level, socioeconomic level, etiology of renal disease, time on dialysis (if applicable), use of medications and the most recent biochemical parameters, no older than 2 months.

Dietary adherence will be measured in patients in the three groups, with a 3-day food consumption record and the application of The renal adherence attitude questionnaire. The level of nutritional knowledge will be measured with the CONURE self-applicable questionnaire, which is a tool to assess knowledge of renal nutrition in dialysis and pre-dialysis patients that was developed and validated (content and appearance) by a group of nutritionists from our hospital. Nutritional status will be assessed by anthropometric measurements (elbow width, weight, height, arm circumference, tricipital skin fold), subjective global assessment or malnutrition inflammation score, protein energy wasting criteria and dynamometry. Finally, quality of life will be assessed with the Kidney Disease Quality of Life - short form 36 (KDQOL-SF36).

The control group will receive standard nutritional care consisting of dietary prescription with follow-up for resolution of doubts and adjustment of the dietary plan every 2-3 months. The intervention group, in addition to the dietary prescription, will receive the educational intervention.

The dietary prescription will be given to the patients of the three groups. Based on the nutritional status, biochemical parameters and stage of renal disease, the dietary plan will be calculated and delivered on the same day as the baseline measurements.

After the initial measurements, the educational intervention will be carried out for the patients in the pre-dialysis group and those in the dialysis group, which will last 5 monthly sessions lasting approximately 2 - 2.5 hours.The content of monthly educational sessions will be: Month 1: proteins (predialysis group), potassium (dialysis group) Month 2: Sodium and fluids (predialysis group), phosphorus (dialysis group) Month 3: Phosphorus (predialysis group), sodium and fluids (dialysis group) Month 4: Potassium (predialysis group), proteins (dialysis group) Month 5: Myths and facts about food (both groups)

Simultaneously to the educational program, in the intervention groups, sessions of a maximum of 5 patients will be held monthly for two hours with a group of clinical psychologists, made up of two people from the center for integral care of patients with diabetes. These sessions will be held on days different from the educational program. In each session the hospital anxiety and depression scale will be applied. The content of the psychological intervention is as follows: Month 1: Psychoeducation with the aim of making participants aware of the psychological aspects of renal disease, grief and the most common barriers to non-adherence to the diet plan, it will facilitate the understanding of the situation they are living and will favor the development of healthy behaviors. Month 2, 3 and 4: Identified barriers will be addressed and, based on this, goals will be established, specifying the behavior to be performed, including frequency, intensity or duration in a given context. In addition, problem-solving therapy will be provided to facilitate active coping that will be useful when facing chronic medical difficulties. Month 5: integrate the relapse prevention strategy, to identify and manage situations that may lead to abandoning new behaviors or adopting new risk behaviors.

After the end of the educational program and the psychological intervention, the patients' records will be reviewed again to extract the most recent biochemical parameters and measurements of dietary adherence, nutritional knowledge, nutritional status and quality of life will be performed for the second time in both the control and intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years old
* Residence in Mexico City, (in order to make it easier for them to attend the educational workshops that will be held within the hospital facilities).
* Patients who are active in the nephrology office of National Institute of Medical Science and Nutrition
* With more than 3 months of diagnosis of chronic kidney disease in pre-dialysis phase (glomerular filtration rate < 60 ml/min/1.73m2) at National Institute of Medical Science and Nutrition
* With more than 3 months with peritoneal dialysis treatment in the National Institute of Medical Science and Nutrition
* With more than 3 months with hemodialysis treatment in the National Institute of Medical Science and Nutrition
* Signed informed consent form

Exclusion Criteria:

* Patients with uncorrected cognitive problems:

  * Patients with post-dialytic syndrome (uremia).
  * Patients with neurological alterations induced by renal failure.
* Patients with mental or psychiatric illness that prevents them from learning and following directions:

  * Patients with persistent delirium
  * Patients with schizophrenia
  * Patients with manic episode
  * Patients with confusional syndrome
  * Patients with minor or major neurocognitive deficits
  * Patients with dissociative amnesia
  * Patients with neurodevelopmental disorder
* Patients who meet Diagnostic and Statistical Manual of Mental Disorders (DSM IV- TR) diagnostic criteria for substance abuse and dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Patients´ dietary attitude | From enrollment to the end of the intervention at 5 months
  Measurement of patients' attitude toward fluid restriction and dietary modifications and their impact on daily life. Adherence to the diet will be measured by the renal adherence attitude questionnaire (RAAQ), at the beginning of the study and after the end of the intervention.
  RAAQ questionnaire will be filled out by the patient with the purpose of evaluating the patients' attitudes and behaviors in relation to diet adherence.
  The questionnaire consists of 26 items with a 5-point Likert scale indicating total agreement (5 points) or total disagreement (1 point). The lowest score on the scale is 26 points and the highest is 130 points. Higher scores on this scale are associated with a more positive patient attitude to dietary restrictions and to a higher dietary adherence.
Dietary adherence | From enrollment to the end of the intervention at 5 months
  Extent to which a patient's eating behavior corresponds to the recommendations agreed upon with the nutritionist. Adherence to the diet will be measured by a three-day food record at the beginning of the study and after the end of the intervention.
  The evaluation of the diet will be carried out by a trained nutritionist, describing the amount and type of food consumed by the patients in a three-day period. The three-day average consumption of calories (kcal), protein (g), sodium, potassium and phosphorus (mg) will be estimated.
  Good adherence will be considered when the actual intake of these nutrients is between 90 and 110% of the recommended intake for each patient.
Nutritional knowledge | From enrollment to the end of the intervention at 5 months
  Assessment of the level of knowledge about food groups and nutrients that are important in chronic kidney disease. Knowledge will be assessed by the CONURE self-administered questionnaire consisting of 35 multiple-choice questions related to sodium, potassium, phosphorus, protein and the use of beverages and nutritional supplements, at the beginning and end of the intervention. The level of knowledge will be classified into three categories according to the number of correct answers obtained: low knowledge with less than 60% correct answers, regular knowledge with 60-80% correct answers and good knowledge with more than 80% correct answers.

SECONDARY OUTCOMES:
Muscle status | From enrollment to the end of the intervention at 5 months
  Measures that quantify a person's muscularity and is a reflection of nutritional status.
  The assessment of muscle status will be performed by calculating the arm muscle area (AMA) which will be compared to the adult reference value (%AMA).
  Patients will be classified as normal muscle status if the %AMA is greater than 90%, as mild, moderate and severe muscle depletion if the %AMA is between 90 and 76%, 75 and 65% and less than 65%, respectively.
Muscle functionality | From enrollment to the end of the intervention at 5 months
  Capacity of muscle mass to perform its functions, mainly related to strength and ability to perform daily activities.
  The measurement of muscle functionality will be performed with dynamometry and is related to the nutritional status of the patients.
  Low strength will be considered when the measurement is < 20 kg in women and < 30 kg in men.
Nutritional status of predialysis patients | From enrollment to the end of the intervention at 5 months
  A person's body situation as a result of the energy balance between caloric intake and metabolic needs. It is an internal condition of the individual that refers to the availability and utilization of energy and nutrients. Nutritional status will be assessed by applying the Subjective Global Score (GSV), which is a diagnostic tool for malnutrition in pre-dialysis patients, before and after the intervention.
  SGA is a tool consisting of 8 questions to which a score between 1 and 7 is assigned according to the alteration of each component. Based on the score obtained, the patient's nutritional status is classified in one of three categories: 1) good nutritional status (6 and 7 points in most of the components), 2) mild/moderate malnutrition (3 to 5 points in most of the components) and 3) severe malnutrition (1 and 2 points in most of the components).
Nutritional status of dialysis patients | From enrollment to the end of the intervention at 5 months
  A person's body situation as a result of the energy balance between caloric intake and metabolic needs. It is an internal condition of the individual that refers to the availability and utilization of energy and nutrients. Nutritional status will be assessed by applying the Malnutrition Inflammation Score (MIS), which is a diagnostic tool for malnutrition in dialysis patients, before and after the intervention.
  MIS is a tool comprising 10 components divided into 4 sections. Each of the evaluated parameters is assigned from 0 to 4 points according to the degree of deficiency. The minimum and maximum score of the tool is 0 and 30 points, respectively.
  The nutritional status is determined according to the sum of the points, with four possible diagnoses: normal nutritional status (< 3 points), mild malnutrition (3 to 5 points), moderate malnutrition (6 to 8 points), severe malnutrition (> 9 points), and severe malnutrition (> 9 points).
Patients´ quality of life | From enrollment to the end of the intervention at 5 months
  Conditions that an individual must enjoy in order to be able to satisfy his needs. This, so that he/she not only survives, but also lives comfortably. The assessment of quality of life will be made at the beginning and end of the intervention, through the self-applicable questionnaire Kidney Disease Quality of Life Short Form (KDQOL-SF36), which consists of a generic section of 12 items related to health status, daily activities and emotional problems, and another specific section of 24 items related to kidney disease, symptomatology and effects of kidney disease on daily life. The response to each of the questions is classified between 1 and up to 6 points according to the degree of affectation. The higher the final score of the questionnaire, the higher the quality of life. Patients will be classified as having good quality of life if they score > 50 points and poor quality of life with < 50 points.

CONTACTS AND LOCATIONS:
Overall Officials: Ximena Atilano Carsi, PhD, Principal Investigator — Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubiránn
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No